CLINICAL TRIAL: NCT00406159
Title: Effects of Hyperbaric Oxygen Therapy on Behavioral Measures of Short Term Memory, Learning, and Behavior in Children With Autism
Brief Title: Effects of Hyperbaric Oxygen Therapy on Children With Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thoughtful House (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06.10.0004
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Autism
Keywords: Autism; Hyperbaric Oxygen Therapy; Behavioral assessments
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy

SUMMARY:
PURPOSE

The purpose of this investigation is to evaluate the cognitive and behavioral effects of Hyperbaric Oxygenation Therapy in children who present with a diagnosis of autism spectrum disorder.

HYPOTHESIS

1. Hyperbaric Oxygenation Therapy will be safe to use with children with autism.
2. Hyperbaric Oxygenation Therapy will have a statistically significant effect on the symptoms of autism.
3. Hyperbaric Oxygenation Therapy will have a clinically significant observable effect on the overt symptoms of autism.
4. The decreases in the symptoms of autism will correlate positively with the number of Hyperbaric Oxygenation Therapy sessions.
5. Treatment gains obtained from Hyperbaric Oxygenation Therapy will be maintained at follow-up, post 40 treatment sessions.

SPECIFIC AIMS

1. Provide further evidence for the safety of Hyperbaric Oxygenation Therapy in children with autism.
2. To quantitatively assess the effects of Hyperbaric Oxygenation Therapy on behavioral and cognitive symptoms of autism before, during, and after treatment.
3. Identify number of treatments required to reach therapeutic effects.
4. Identify the length and durability of treatment effect and maintenance.

DETAILED DESCRIPTION:
Participants & Setting

Participants in this study will be 30 consecutive children referred to Thoughtful House for the treatment of autism or a related developmental disorder. Participants may or may not also be concurrently receiving intensive behavioral intervention services from the Center for Autism and Related Disorders. All therapy and behavioral testing sessions will occur on the premises of Thoughtful House.

Inclusion Criteria

The following criteria will be considered inclusionary:

* Male and female children 2-10 years diagnosed with autism, PDD, or Aspergers
* No anticipated changes in treatment for the study duration (e.g., diet, nutrients)

  * No additional biomedical treatments started 6 weeks prior to enrollment
  * No changes in dietary management for 3 months prior to enrollment
* Access to Thoughtful House on a daily basis, or as necessary for the study participation

In addition, the child participant must be:

* Ambulatory or require minimum support walking, per parent
* Able to sit still for 5 minutes or longer with a preferred toy item, per parent
* Adequate vision and hearing for the purposes of test administration, per parent
* Adequate arm-hand-finger coordination (i.e., able to point) for learning and cognitive tasks used in outcome measurement, per parent
* Stable and controlled medical disorder
* Under the care of a caregiver willing to participate by attending regularly scheduled appointments and completing the necessary measures

Exclusion criteria

The following criteria will be considered exclusionary:

Current otitis media Sinus infection Asthma Pulmonary cysts Emphysema Upper respiratory infection Severe claustrophobia, intolerance to being in the chamber History of Seizures Unstable/uncontrolled disorder of any kind

Design Ten sets of multiple baseline measurement groups, 3 participants each (n=30) will be used to evaluate the effects of HBOT on the behavioral measures of adaptive (mean length of utterance, MLU), aberrant, and stereotyped behaviors. The first participant in each multiple baseline will receive sessions of the behavioral measures for a minimum of one week prior to the implementation of HBOT. Subsequent participants cannot receive HBOT until an effect is observed (as determined via visual inspection and statistical analysis of the data) on prior participants or until prior participants have received 40 HBOT treatments, whatever occurs first. Subsequent to receiving 40 HBOT treatments, each participant will be given a break from HBOT for at least one week, during which time the schedule of behavioral measures will remain the same. If proficiency on the behavioral measures decreases when HBOT is terminated for one week, HBOT may be reinitiated as per the discretion of the physician and parent.

HBOT Systematic Desensitization

Because children with autism often do not tolerate changes in the environment, we anticipate difficulties with initial treatment compliance in some children. In a clinical setting, children become acquainted with the mask and machine, and are introduced to an enclosed oxygen chamber and HBOT begins at a prescribed pressure. Below are the general desensitization procedures for the participants:

1. The child is introduced to the mask and therapist models how it is worn
2. The child is required to hold the un-strapped mask loosely against his/her face until he/she can breathe while holding the mask in place for a minute or more
3. The child is required to strap the mask on for a minute, with gradual increase to 30+ minutes
4. The child is seated upright in the chamber with the mask on and the HBOT machine off for a minute, with a gradual increase to 30+ minutes
5. The child is lying down in the chamber with the mask on and the HBOT machine on at a low pressure setting for a minute, with gradual increase to 30+ minutes
6. The child has the mask strapped on and lying down, while the HBOT is running for an hour

For some children who exhibit severe noncompliance with the HBOT procedure, relaxation training and listening to preferred music prior to the HBOT procedure may be used.

In order to minimize the influence of learning and attention from parents/therapists during HBOT/placebo sessions, all children will be viewing a developmentally-appropriate DVD (e.g., Disney movie) during all HBOT sessions to minimize confounding effects that may occur with other activities. The viewing of DVDs will continue throughout all 80 sessions and during follow-up.

Procedures Data will be collected according to the following schedule: prior to treatment, following 5, 15, 25, and 40 HBOT treatments, as well as at post-treatment and 1 and 3-month follow-up.

Behavioral Measures Participants who are receiving intensive behavioral intervention services during the course of the study will have continuous measures of many aspects of performance recorded daily, as a part of their behavioral intervention services. Such measures will be customized to the behavioral education needs of each child, but are likely to include, at a minimum: 1) measure of adaptive behavior (e.g., language); 2) measure of aberrant behavior (e.g., tantrums, etc.); and 3) stereotyped behavior. All such continuous measures can be observed throughout the course of the participant's involvement in the study. However, the consideration of any particular continuous measure as part of the current study would require inter-observer agreement data be collected on those measures for a minimum of 25% of the observed data. That is, a second, independent observer must record data on all behavioral clinical measures which will be included in the study. Participants who are not receiving intensive behavioral intervention services will receive only the behavioral measures described below. Participants who are receiving intensive behavioral intervention services during the course of the study will receive the measures described below, as well as any of their clinical behavioral measures for which adequate inter-observer agreement data are collected.

Repeated acquisition task

A defining feature of autism is a global impairment in one's ability to learn. Repeated acquisition tasks are commonly used in drug behavioral pharmacology studies to assess the effect of a drug on the ability of an individual to learn, that is, the efficiency with which the individual's behavior is brought under new forms of stimulus control. Repeated acquisition tasks typically involve the participant learning to respond to a new sequence of positions during each session. For example, four levers or buttons are presented and the participant must press the four buttons in a particular sequence in order to earn reinforcement. However, the correct sequence is different for every session, and typically one session is conducted daily, so the sequence of responding required to earn reinforcement is different each day. The performance of the participant can be analyzed in a number of ways including the percent correct for the entire session, the total number of responses or the number of errors made until 80% correct responding is reached.

The complexity of the task can be adjusted by varying either or both of two parameters: 1) the number of response positions present (e.g., number of buttons present), and 2) the number of responses in the sequence required for reinforcement. For example, ten buttons could be present but the participant is only required to press one particular button out of the ten in order to get reinforcement, versus pressing a sequence of ten which involves each button once, versus having only two buttons present, etc. The standard degree of complexity in behavioral pharmacology research is having four response options present and requiring the participant to respond to all four in a particular order to earn reinforcement.

Delayed matching to sample

An additional cognitive process that might be of interest when evaluating HBOT is short-term memory. A common behavioral measure of short-term memory is a delayed matching-to-sample (DMTS) procedure. In such procedures, a sample stimulus is presented and then removed and a delay occurs between the removal of the sample stimulus and the presentation of two or more comparison stimuli. The participant earns reinforcement for choosing the correct comparison stimulus. The delay between the removal of the sample stimulus and the presentation of the comparison stimuli can vary from zero to any conceivable duration, but typically does not exceed 60 seconds.

The relation between the sample stimulus and the correct comparison stimulus can be varied in order to alter the difficulty of the task. For example, the sample stimulus and the correct comparison stimulus may be identical, often referred to as "identity matching." This is the easiest form of DMTS. Alternatively, the sample stimulus may be related to the correct comparison stimulus in an abstract dimension. For example, the sample stimulus may be the written word car and the correct comparison stimulus might be a bicycle, with a gorilla and a fork as distracters.

Sessions can be conducted with a fixed delay or the delay can be systematically increased during the session in order to identify a threshold at which the participant is no longer able to respond correctly. For example, on the first trial, the delay may be zero second and then the delay may be increased by 4 seconds on each subsequent trial, contingent on correct responsse on the previous trial. The data are then analyzed to determine the longest delay at which the participant was consistently correct at 80% accuracy. This threshold can be considered a measure of the participant's short term memory at the time of the session.

Standardized Measures

In addition to the direct measures of behavior described above, standardized intelligence and adaptive assessments will be conducted prior to the initiation of HBOT. These will include:

ADI/ADOS WPPSI-III (2-6 years) /WASI (6+ years) Vineland Adaptive Behavior Scale (VABS) Subjective Questionnaires Aberrant Behavior Checklist Clinical Global Impression ATEC Selected sections of the APEQ BRIEF Parenting Stress Index Repetitive Behavior Scale A side effect questionnaire Thoughtful House Caregiver diary

Laboratory & Physiological Measures Full physical exam (weight, height, vital signs-temperature) Otoscopic examination prior to enrollment in the study

STATISTICAL DESIGN/ANALYSIS

The primary measures will consist of changes in the rate and percentage of change from pre and post HBOT adaptive, aberrant, and stereotyped behaviors.

ADVERSE EFFECTS AND MANAGEMENT: the only 2 most commonly encountered adverse reactions are ear pain and sinus pressure.

Ear Pain: This can be minimized or ameliorated by working on pressure equalization techniques across the tympanic membrane. These techniques include:

Yawning Drinking water/juice Val Salva (Plugging nose and mouth, blowing air out the ears) Jaw thrust and swallowing Bending head to the side and yawning/swallowing. The technician can slow the rate of pressurization allowing adequate time for pressure equalization to occur

Sinus pressure: this can be ameliorated with slowing down the rate of pressurization and depressurization. Also, the administration of 0.5% Neosynephrine intranasally and pseudoephedrine can be used.

Should a serious adverse event occur, the form SERIOUS ADVERSE EVENT REPORTING FORM will be filled out and reported to the IRB office within 5 business days and a written summary of the circumstances surrounding the adverse reaction be submitted to the IRB for review at the next scheduled IRB meeting.

Minor reactions, such as ear pain or sinus pressure will be managed and documented by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children 2-10 years diagnosed with autism, PDD, or Aspergers
* No anticipated changes in treatment for the study duration (e.g., diet, nutrients)
* No additional biomedical treatments started 6 weeks prior to enrollment
* No changes in dietary management for 3 months prior to enrollment
* Access to Thoughtful House on a daily basis, or as necessary for the study participation
* In addition, the child participant must be:

  * Ambulatory or require minimum support walking, per parent
  * Able to sit still for 5 minutes or longer with a preferred toy item, per parent
  * Adequate vision and hearing for the purposes of test administration, per parent
  * Adequate arm-hand-finger coordination (i.e., able to point) for learning and cognitive tasks used in outcome measurement, per parent
  * Stable and controlled medical disorder
  * Under the care of a caregiver willing to participate by attending regularly scheduled appointments and completing the necessary measures

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Standardized Measures
In addition to the direct measures of behavior described above, standardized intelligence and adaptive assessments will be conducted prior to the initiation of HBOT. These will include:
ADI/ADOS
WPPSI-III (2-6 years) /WASI (6+ years)
Vineland Adaptive Behavior Scale (VABS)
Subjective Questionnaires
Aberrant Behavior Checklist
Clinical Global Impression
ATEC
Selected sections of the APEQ
BRIEF
Parenting Stress Index
Repetitive Behavior Scale
A side effect questionnaire
Thoughtful House Caregiver diary

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wakefield, MD, Study Director — Thoughtful House Center for Children
Locations (1):
- Medical Center at Thoughtful House, Austin, Texas, United States

REFERENCES:
- [Result] Rossignol DA, Rossignol LW. Hyperbaric oxygen therapy may improve symptoms in autistic children. Med Hypotheses. 2006;67(2):216-28. doi: 10.1016/j.mehy.2006.02.009. Epub 2006 Mar 22. PMID 16554123
- [Derived] Jepson B, Granpeesheh D, Tarbox J, Olive ML, Stott C, Braud S, Yoo JH, Wakefield A, Allen MS. Controlled evaluation of the effects of hyperbaric oxygen therapy on the behavior of 16 children with autism spectrum disorders. J Autism Dev Disord. 2011 May;41(5):575-88. doi: 10.1007/s10803-010-1075-y. PMID 20680427